CLINICAL TRIAL: NCT00002430
Title: A Multicenter, Open-Label, 24-Week Study to Compare the Safety and Activity of Indinavir Sulfate/d4T/3TC Versus Indinavir Sulfate/Nelfinavir Mesylate/d4T/3TC in HIV-Infected Individuals
Brief Title: A Study to Compare the Effectiveness of Two Anti-HIV Drug Combinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 246R; 079-02; CRX454
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-02

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Lamivudine; Indinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Nelfinavir
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Nelfinavir; Lamivudine; Stavudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Nelfinavir mesylate
Drug: Lamivudine
Drug: Stavudine

SUMMARY:
The purpose of this study is to compare two different anti-HIV drug combinations, one that contains nelfinavir (NFV) and one that does not. The best dosing schedule for indinavir (IDV) also will be studied.

DETAILED DESCRIPTION:
Patients are stratified by screening plasma viral RNA results (50,000 copies/ml or below vs above 50,000 copies/ml) and randomized to 1 of 2 treatment arms. Group 1 receives IDV 3 times daily plus d4T/3TC twice daily. Group 2 receives IDV/NFV/d4T/3TC twice daily. Patients remain on study medications for 24 weeks and are seen at the clinic once every 4 weeks after entering the study. At each clinic visit, blood samples are taken to evaluate CD4 cell count and plasma HIV RNA levels.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV positive.
* Have a viral load (level of HIV in your blood) of at least 10,000 copies/ml within 45 days of study entry.
* Have a CD4 cell count of at least 100 cells/mm3 within 45 days of study entry.
* Have a normal chest X-ray.
* Have never taken protease inhibitors or 3TC.
* Are 16 years of age or older.
* Agree to practice sexual abstinence or use barrier methods of birth control (e.g., condoms).

Exclusion Criteria

You will not be eligible for this study if you:

* Have an active opportunistic (AIDS-related) infection or cancer.
* Have certain types of Kaposi's sarcoma.
* Have hepatitis.
* Have chronic diarrhea.
* Have a history of certain medical conditions.
* Are allergic to any of the study medications.
* Are taking certain medications.
* Are pregnant or breast-feeding.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220

CONTACTS AND LOCATIONS:
Locations (46):
- United States (46):
  - Univ of Alabama School of Med, Montgomery, Alabama
  - Ocean View Internal Medicine, Long Beach, California
  - AIDS Healthcare Foundation, Los Angeles, California
  - Tower ID Med Associates, Los Angeles, California
  - Oasis Clinic / King Drew Med Ctr, Los Angeles, California
  - Robert Scott MD, Oakland, California
  - AIDS Community Research Consortium, Redwood City, California
  - Saint Francis Mem Hosp / HIV Care Unit, San Francisco, California
  - Pacific Horizons Med Group, San Francisco, California
  - Kaiser Foundation Hospital, San Francisco, California
  - Harbor - UCLA Med Ctr, Torrance, California
  - Denver Public Health Dept, Denver, Colorado
  - Blick Med Associates, Stamford, Connecticut
  - Physicans Home Service, Washington D.C., District of Columbia
  - IDC Research Initiative, Altamonte Springs, Florida
  - Univ of Miami School of Medicine, Miami, Florida
  - Hillsborough County Health Dept, Tampa, Florida
  - Emory Univ, Atlanta, Georgia
  - Harold Katner MD, Macon, Georgia
  - Thomas Coffman MD, Boise, Idaho
  - Chicago Ctr for Clinical Research, Chicago, Illinois
  - Northwestern Univ Med Ctr, Chicago, Illinois
  - Univ of Illinois, Chicago, Illinois
  - Kentucky Clinical Research, Lexington, Kentucky
  - Louisiana State Univ Med Ctr / Tulane Med School, New Orleans, Louisiana
  - AIDS Consultation Service / Maine Med Ctr, Portland, Maine
  - Institute of Human Virology, Baltimore, Maryland
  - JSI Research and Training Institute, Boston, Massachusetts
  - Education & Research Building, Camden, New Jersey
  - NJCRI, Newark, New Jersey
  - Infectious Disease Specialists of NJ, Union, New Jersey
  - Brookdale Univ Hosp and Med Ctr, Brooklyn, New York
  - Liberty Med Group, New York, New York
  - James Jones MD, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Community Health Network, Rochester, New York
  - Wake Forest Univ School of Medicine, Winston-Salem, North Carolina
  - Associates in Med and Mental Health, Tulsa, Oklahoma
  - The Research and Education Group, Portland, Oregon
  - Fanno Creek Clinic, Portland, Oregon
  - Anderson Clinical Research / Inc, Pittsburgh, Pennsylvania
  - Burnside Clinic, Columbia, South Carolina
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Oak Lawn Physicians Group, Dallas, Texas
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Infections Ltd / Physicians Med Ctr, Tacoma, Washington